CLINICAL TRIAL: NCT03331107
Title: Correlation of the Objective and Subjective Measures of the Nasal Obstruction Before and After Surgery of the Nasal Septum
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SEPTORHINO
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nasal obstruction is a very subjective sensation but it's also a frequent reason of consultation. Two specific questionnaire NOSE and RhinoQOL were validated; but rhinomanometry value is still a question to debate. As well as the difference between acoustic rhinometry and rhinomanometry.

Usually nasal obstruction due to a septal deviation is treated by septoplasty. If the anatomic result can be proved true, the patient's felt would be unsuccessful.

The aim of this study is to assess the impact of septoplasty on the nasal obstruction, objectively by rhinometry and subjectively by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* with medical insurance
* programmed for septoplasty
* nasal obstruction with septal deviation
* accept participation

Exclusion Criteria:

* nasal sine polyposis
* endonasal mass
* chronic sinusite
* previous nasal surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient admitted for septoplasty in Institut Arthur Vernes
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Nose Obstruction symptom Evaluation | 3 months
  scale about nose obstruction filled up by the patient
nasal resistance to airflow | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France